CLINICAL TRIAL: NCT01502540
Title: Pain Prevalence After Major Craniotomy in Siriraj Hospital
Brief Title: Pain Prevalence After Major Craniotomy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Other Study IDs: Si223/2011; 161/2554(EC1) (Other: Faculty of Medicine, Siriraj Hospital)
Record Dates: First submitted 2011-12-29; First posted 2011-12-30 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Pain; Craniotomy
Keywords: pain; craniotomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Craniotomies are generally thought to be less painful than other operations. Indeed recent studies have confirmed that pain is a common problem during the postoperative phase following craniotomy.Pain not only causes discomfort, but it is also associated with other potential adverse events such as increased sympathetic activity and elevated systemic blood pressure. These events in turn may contribute to increased intracranial pressure. Some patients may also develop chronic pain.Potent opioids have been avoided due to its potential to cause respiratory depression and risk of masking pupillary signs. As a result postoperative craniotomy pain controls are usually inadequate.

In Siriraj hospital, there are 500-600 craniotomy patients per year. Still there are no definite guidelines for postoperative pain management in these patents due to lack of information about quality of postoperative pain control after craniotomy.

Objectives

Primary objective :

- To study incidence of moderate to severe pain during first 48 hours after craniotomy.

Secondary objectives :

* To determine risk factors for moderate to severe pain during first 48 hours after craniotomy
* To evaluate side effects and complications of postoperative craniotomy pain control
* To compare patient's expectation for pain management before and after surgery
* To determine patient's satisfaction for postoperative pain management

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing major craniotomy (supratentorial surgery and Infratentorial surgery)
* Age > 18 years

Exclusion Criteria:

* Emergency or trauma
* Need postoperative ventilatory support
* Cannot communication
* Psychosis
* Not adherence to the treatment protocol
* History of using benzodiazepine or addictive substance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing cranitomy
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
incidence of moderate to severe pain following major craniotomy | 48 hours

SECONDARY OUTCOMES:
risk factors of moderate to severe pain following craniotomy. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Sirilak Suksompong, Bangkok, Thailand